CLINICAL TRIAL: NCT06196879
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multi-center, Dose-ranging Study to Evaluate the Efficacy and Safety of Verekitug (UPB-101) in Adult Participants With Severe Asthma (VALIANT)
Brief Title: A Study to Investigate the Efficacy and Safety of Verekitug (UPB-101) in Adult Participants With Severe Asthma (VALIANT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Upstream Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPB-CP-04; 2023-507410-27-00 (Other: EUCT)
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Severe Asthma
Keywords: VALIANT; Respiratory Tract Diseases; Bronchial Diseases; Asthma; Lung Diseases; Uncontrolled Asthma; Severe Asthma
MeSH Terms: conditions — Asthma; Respiratory Tract Diseases; Bronchial Diseases; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Verekitug (UPB-101): 100 mg Q12W / Placebo (Experimental): Participants will receive 0.5 milliliter (mL) of verekitug (UPB-101) formulated solution (containing 100 milligrams [mg] of verekitug [UPB-101]) and 2.0 mL of placebo subcutaneously in two separate injections every 12 weeks up to Week 48.
  Interventions: Drug: Verekitug (UPB-101); Drug: Placebo
- Verekitug (UPB-101): 400 mg Q24W / Placebo (Experimental): Participants will receive 2.0 mL of verekitug (UPB-101) formulated solution (containing 400 mg of verekitug [UPB-101]) and 0.5 mL of placebo subcutaneously in two separate injections every 24 weeks up to Week 48. Participants will also receive 2 mL and 0.5 mL of placebo subcutaneously in two separate injections at Weeks 12 and 36 visits.
  Interventions: Drug: Verekitug (UPB-101); Drug: Placebo
- Verekitug (UPB-101): 100 mg Q24W / Placebo (Experimental): Participants will receive 0.5 mL of verekitug (UPB-101) formulated solution (containing 100 mg of verekitug [UPB-101]) and 2.0 mL of placebo subcutaneously in two separate injections every 24 weeks up to Week 48. Participants will also receive 2 mL and 0.5 mL of placebo subcutaneously in two separate injections at Weeks 12 and 36 visits.
  Interventions: Drug: Verekitug (UPB-101); Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive 0.5 mL of matching placebo and 2.0 mL of matching placebo subcutaneously in two separate injections every 12 weeks up to Week 48.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verekitug (UPB-101) — Verekitug (UPB-101) formulated solution
  Arms: Verekitug (UPB-101): 100 mg Q12W / Placebo; Verekitug (UPB-101): 100 mg Q24W / Placebo; Verekitug (UPB-101): 400 mg Q24W / Placebo
Drug: Placebo — Verekitug (UPB-101) matching placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of verekitug (UPB-101) in participants with severe asthma. The study will evaluate the incidence of asthma exacerbations, other pharmacodynamic (PD) parameters such as lung function and asthma control, and the safety and tolerability of verekitug (UPB-101) compared to placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled, parallel group study to assess the efficacy and safety of verekitug (UPB-101) administered subcutaneously (SC). A total of approximately 436 adult participants with severe asthma are planned for enrolment and will be randomized in a 1:1:1:1 ratio to receive verekitug (UPB-101) at doses of 100 mg every 12 weeks (Q12W), 400 mg every 24 weeks (Q24W), and 100 mg every 24 weeks (Q24W), or placebo administered SC. In order to maintain the blinding of different doses, all participants will receive 2 SC injections at each dosing visit. This study consists of a Screening/Run-In Period (approximately 4 weeks), Treatment Period (up to 60 weeks with a minimum of 24 weeks) and Follow-up Period (ending approximately 16 weeks after the last administration of study intervention).

ELIGIBILITY:
Inclusion Criteria:

* Signed, dated, and received a copy of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent form (ICF).
* Age 18 to 80 years of age (inclusive) at the time of consent.
* Physician-diagnosed asthma for at least 12 months prior to Visit 1.
* Participant has evidence of bronchodilator (BD) reversibility as documented by either historical reversibility (within 12 months prior to study entry) or reversibility during screening.
* Documented treatment with a total daily dose of either medium or high dose inhaled corticosteroids (ICS) for at least 3 months. Participants on medium dose ICS must also have been taking at least one additional maintenance asthma controller medication for at least 3 months.
* Documented history of asthma exacerbation(s) within 12 months of Visit 1.
* Asthma Control Questionnaire-6 (ACQ-6) score greater than or equal to (>=) 1.5 at screening and randomization.
* Participant must have a pre-BD FEV1 value of >=30 percent (%) and <=80% predicted at Screening.
* Minimum compliance with daily diary and background asthma medication(s) as captured in the daily diary during the Run-in Period.
* Agrees to follow the required contraceptive techniques/methods.
* Female or male participant agrees not to donate eggs or sperm, respectively, for a period of 120 days after the last dose of the study drug intervention or at the Final Visit, whichever occurs last.

Exclusion Criteria:

* Inpatient hospitalization due to asthma at any time within 4 weeks prior to Visit 1 or during the Screening/Run-in Period.
* Previous exposure to verekitug (UPB-101) or known allergy/sensitivity to any of its excipients.
* Previous biologics, including those for asthma treatment, for which the appropriate washout period is not fulfilled prior to Visit 1. If the half-life is not known, a 24-week washout period prior to Visit 1 should be applied.
* Allergen immunotherapy (unless maintenance dose) within 12 weeks prior to Visit 1 or plans to begin therapy or change dosing during the study.
* For participants taking oral corticosteroids (OCS), the dose has not been stable for at least 2 weeks prior to Visit 1 and/or is >10 milligram (mg) daily, or >20 mg every other day.
* Evidence of active or suspected bacterial, viral, fungal, or parasitic infections within 2 weeks prior to Visit 1.
* History compatible with or diagnosis of a parasitic infection and has not been treated or has not responded to standard of care therapy.
* Current tobacco smokers, nicotine vapers (including electronic cigarettes), snuff users or participants with a smoking history >=10 pack years. (Former nicotine smokers with a smoking history of <10 pack years, former nicotine vapers and former snuff users must have stopped for at least 6 months prior to Visit 1 to be eligible).
* Positive coronavirus disease 2019 (COVID-19) test with lower respiratory tract symptoms within 28 days before Visit 1.
* Pregnant or breastfeeding or planning to become pregnant or breastfeed during the study or unwilling to use adequate birth control, if of reproductive potential and sexually active.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Annual Asthma Exacerbation Rate (AAER) | Baseline up to Week 60
  An asthma exacerbation is defined as a worsening of asthma that required treatment with systemic (oral or intravenous) corticosteroids for at least three consecutive days or a single depo-injectable dose of corticosteroids or an emergency room (ER) or urgent care visit that required systemic corticosteroids or an admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for greater than or equal to 24 hours.

SECONDARY OUTCOMES:
Change from Baseline in Forced Expiratory Volume in 1 Second (FEV1) of Pre-bronchodilator (Pre-BD) to Week 60 | Baseline to Week 60
  Spirometry will be performed pre-bronchodilator (BD) to measure lung function. FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Change from Baseline in Fractional exhaled nitric oxide (FeNO) to Week 60 | Baseline to Week 60
  Standardized single breath FeNO test is performed to evaluate airway inflammation.
Change from Baseline in Asthma Control Questionnaire-6 (ACQ-6) to Week 60 | Baseline to Week 60
  ACQ-6 is a participant-reported questionnaire to assess asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs | Up to Week 64
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: James C Lee, MD, Study Director — Upstream Bio
Locations (155):
- United States (55):
  - AllerVie Clinical Research, Birmingham, Alabama
  - Kern Research, Inc., Bakersfield, California
  - Velocity Clinical Research - Lafayette LA, Los Angeles, California
  - Newport Native MD Inc, Newport Beach, California
  - California Medical Research Associates Inc., Northridge, California
  - Integrated Research of Inland Inc, Upland, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Allianz Research Institute, Westminster, California
  - Woodland Clinic Medical Group, Woodland, California
  - National Jewish Health, Denver, Colorado
  - Advance Pharma Research, Cutler Bay, Florida
  - Unique Clinical Trials, Doral, Florida
  - Health and Life Research Institute, LLC, Miami, Florida
  - Phoenix Medical Research, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Nouvelle Clinical Research, Miami, Florida
  - Anderson Allergy And Asthma, PA, Orlando, Florida
  - Edward Jenner Research Group, LLC, Plantation, Florida
  - R&B Medical Center, Tampa, Florida
  - Clinical Site Partners dba Flourish research, Winter Park, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Pivotal Research Solutions, Stonecrest, Georgia
  - RNA America Health Sciences, Sugar Hill, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Velocity Clinical Research - Meridian, Meridian, Idaho
  - Howard County Center for Lung and Sleep Medicine LLC, Columbia, Maryland
  - Chesapeake Clinical Research Inc, White Marsh, Maryland
  - Exordia Medical Research Inc, Fall River, Massachusetts
  - Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan
  - AA Medical Research Center, Flint, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - M3 Wake Research, Las Vegas, Nevada
  - Urban Health Plan INC, The Bronx, New York
  - Advanced Respiratory and Sleep Medicine LLC, Huntersville, North Carolina
  - Summit Research Group LLC, Munroe Falls, Ohio
  - Toledo Institute of Clinical Research Inc, Toledo, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Portland Clinical Research, Clackamas, Oregon
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - WR-Notus Clinical Research, LLC, Charleston, South Carolina
  - Velocity Clinical Research - Spartanburg, Spartanburg, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Horizon Clinical Research, Cypress, Texas
  - Alina Clinical Trials, LLC, Dallas, Texas
  - AARA Research Center, Dallas, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - Greater Houston Memorial Pulmonary and Sleep, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Mayflower Clinical, Marble Falls, Texas
  - Metroplex Pulmonary and Sleep Center Drive, McKinney, Texas
  - Element Research Group, San Antonio, Texas
  - DM Clinical Tomball, Tomball, Texas
  - Velocity Clinical Research, West Jordan, Utah
  - University of Wisconsin--Madison, Madison, Wisconsin
- Argentina (14):
  - CARE: Centro de Alergia y Enfermedades Respiratorias, Buenos Aires, Argentina
  - Fundacion Respirar - Centro Medico Dra. De Salvo, Buenos Aires, Argentina
  - Fundacion Cidea, Caba, Argentina
  - InAER, CABA, Argentina
  - Centro Medico Dharma, Mendoza, Argentina
  - IERIM Instituto de Enfermedades Respiratorias e Investigacion Medica, San Juan Bautista, Buenos Aires
  - Centro Dr. Lazaro Langer Privado Medicina del Aparato Respiratorio, Córdoba, Córdoba Province
  - Centro de Medicina Respiratoria, Concepción del Uruguay, Entre Ríos Province
  - Fundacion Scherbovsky, Mendoza, Mendoza Province
  - INSARES, Mendoza, Mendoza Province
  - Fundacion Estudios Clinicos (FECLIN), Rosario, Santa Fe Province
  - Instituto Especialidades de la Salud Rosario, Rosario, Santa Fe Province
  - Office of Hector H. Altieri MD, San Miguel de Tucumán, Tucumán Province
  - Investigaciones En Patologias Respiratorias, San Miguel de Tucumán, Tucumán Province
- Bulgaria (10):
  - MHAT "Rahila Angelova" Pernik, Pernik, Pernik
  - UMHAT Sveti Georgi, Plovdiv, Plovdiv
  - Ambulatory For Specialized Outpatient Medical Care - Individual Practice - Dr. Nikolay Evgeniev Ruse Ltd, Rousse, Ruse
  - Medical Center Excelsior, Sofia, Sofia
  - Medical Center HERA EOOD, Sofia, Sofia
  - DCC Convex, Sofia, Sofia
  - Medconsult Pleven, Sofia, Sofia
  - Medical center Pulmovizhyn, Sofia, Sofia
  - Medical Center New Rehabilitation Center EOOD, Stara Zagora, Stara Zagora
  - MC Zdrave 1, Vratsa, Vratsa
- Canada (4):
  - Dynamic Drug Advancement, Ajax, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Toronto Allergists, Toronto, Ontario
  - Winchester Hospital, Winchester, Ontario
- Chile (5):
  - Centro Médico BIOREUMA, Concepción, Chile
  - CIMER, Providencia, Chile
  - Sociedad medica Sy G Limitada, Santiago, Chile
  - Fundacion Medica San Cristobal, Santiago, Santiago Metropolitan
  - Icegclinic, Santiago, Santiago Metropolitan
- Czechia (4):
  - Fakultni Nemocnice u Sv. Anny v Brne, Brno, Czech Republic
  - Alergologie a imunologie Hofstetr Alois MUDr. s.r.o., Jihlava, Czech Republic
  - Plicni Stredisko Teplice S.R.O, Teplice, Czech Republic
  - PNEUMOLOGIE VARNSDORF s.r.o., Varnsdorf, Czech Republic
- Germany (8):
  - IKF Pneumologie Frankfurt, Clinical Research Center Respiratory Diseases, Hessen, Germany
  - IKF Pneumologie GmbH & Co. KG, Mainz, Germany
  - ME Clinical Respiratory Research Hamburg GmbH, Hamburg, Hamburg
  - KPPK Studienzentrum, Koblenz, Rhineland-Palatinate
  - POIS Sachsen GmbH, Leipzig, Saxony
  - RCMS/Lungenpraxis Hohenzollerndamm, Berlin, State of Berlin
  - Velocity Clinical Research Germany , Berlin, Berlin, State of Berlin
  - Pneumologisches Studienzentrum, Berlin, State of Berlin
- Italy (4):
  - Ospedale San Martino, Genova, Genova
  - UOSD Allergologia e Immunodeficienze dell'A.O.U. Federico II, Napoli, Napoli
  - Fondazione IRCCS Policlinico "San Matteo" - SC Pneumologia', Pavia, Pavia
  - SSD Asma Grave e Malattie Rare del Polmone, AOU San Luigi Gonzaga, Orbassano, Torino
- Japan (9):
  - KKR Sapporo Medical Center, Sapporo, Hokkaido
  - Oji General Hospital, Tomakomai, Hokkaido
  - National Hospital Organization Ibarakihigashi National Hospital, Ibaraki, Ibaraki
  - Osaka Metropolitan University Hospital, Osaka, Japan
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Kishiwada City Hospital, Kishiwada, Osaka
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinics, Chuo-ku, Tokyo
- Poland (12):
  - Centrum Badan Klinicznych, Wroclaw, Dolnoslaskie Voivodeship
  - "ALL-MED" Specjalistyczna Opieka Medyczna. Medyczny Instytut Badawczy, Wroclaw, Dolnoslaskie Voivodeship
  - Lekarze Specjalisci - J. Malolepszy I Partnerzy, Wroclaw, Dolnoslaskie Voivodeship
  - Centrum Medyczne All-Med Spolka Komandytowa, Krakow, Malopolskie Voivodeship
  - Nzoz Atopia, Krakow, Malopolskie Voivodeship
  - Malopolskie Centrum Alergologii, Krakow, Malopolskie Voivodeship
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp Z O.O., Tarnów, Malopolskie Voivodeship
  - Prywatny Gabinet Lekarski Malgorzata Pawlukiewicz, Rzeszów, Podkarpackie Voivodeship
  - EMED Centrum Uslug Medycznych, Rzeszów, Podkarpackie Voivodeship
  - Centrum Medycyny Oddechowej, Mroz Spolka Jawna, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Klinika Alergologii i Pneumonologii, Gdansk, Pomorskie Voivodeship
  - Ostrowieckie Centrum Medyczne spolka cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- South Africa (6):
  - Synapta Clinical Research Centre, Durban, Durban
  - Newtown Clinical Research Centre, Johannesburg, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - St Augustine's Hospital/Dr. IA Abdullah, Durban, KwaZulu-Natal
  - University of Cape Town Lung Institute, Cape Town, Western Cape
- South Korea (10):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Bucheon
  - Chungbuk National University Hospital, Cheongju-si, Chubgbuk
  - Yeungnam University Hospital, Daegu, Daegu
  - Eunpyeong St. Marys Hospital, Seoul, Korea
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul, Republic of Korea
  - Asan Medical Center, Seoul, Seoul
  - Kyung Hee University Hospital, Seoul, Seoul
  - Seoul National University Hospital, Seoul, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
- Spain (2):
  - Giromed Institute, Girona, Barcelona
  - Hospital Gregorio Marañon, Madrid, Madrid
- Ukraine (3):
  - Chernivtsi Regional Clinical Hospital, Chernivtsi, Chernivtsi Oblast
  - Municipal non-Profit Enterprise "lvano-Frankivsk Regional Phthisiology-Pulmonology Center of lvano-Frankivsk regional council, Ivano-Frankivsk, Ivano-Frankivs'k
  - Medical Centre "Neuromed" of Limited Liability Company "Scan Light", Vinnytsia, Vinnytsia Oblast
- United Kingdom (9):
  - Hull University Teaching Hospitals NHS Trust, Cottingham, East Yorkshire
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - Ormeau Clinical Trials Ltd, Belfast, Northern Ireland
  - Churchill Hospital, Oxford, Oxfordshire
  - Asthma/COPD Clinical Research Centre, Glasgow, Scotland
  - St Peter's Hospital, Chertsey, Surrey
  - Heartlands Hospital, University Hospitals Birmingham NHS Trust, Birmingham, West Midlands
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Duckworth Lane Clinical Research Facility, Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: No